CLINICAL TRIAL: NCT03770650
Title: Comparison of Intravascular Ultrasound-guided With Angiography-guided Double Kissing Crush Stenting Technique for Patients With Complex Coronary Bifurcation Lesions: The Prospective, Multi-center, Randomized DKCRUSH VIII Trial
Brief Title: IVUS-guided DK Crush Stenting Technique for Patients With Complex Bifurcation Lesions
Acronym: DKCRUSH-VIII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Shaoliang Chen, MD, Vice President, Nanjing First Hospital, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFH20180920
Record Dates: First submitted 2018-12-06; First posted 2018-12-10 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Intervention Model Description: Patients will undergo 1:1 randomization to either IVUS-guided DKCrush stenting which will be the treatment group or Angio-guided DKCrush stenting which will be the control group based on an online Clinical Research Data Management Platform provided by King Yee,,Beijing CN. The initiation of the trial is defined as the time of randomization. After study subjects' enrollment and randomization, the study intervention will take place immediately. The follow-up visits for the primary endpoint are scheduled at 1, 6, and 12 months after the index procedure. Angiographic follow-up is scheduled at 13 months.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will remain blinded until the final study results are released.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IVUS-guided DK crush stenting (Experimental): In the IVUS-guided DK crush stenting group, IVUS will be before side branch stenting, after rewiring side branch, after 1st kissing balloon inflation, after rewiring side branch, after 2nd kissing balloon inflation.
  For LM bifurcation lesions involving ostial LAD and LCX: minimum stent are (MSA) should be ≥10mm2 (LM), 7 mm2 (LAD), and 6 mm2 (LCX), with stent expansion index ≥90% (CSA≥90% of distal reference lumen area in LCX) and symmetry index >0.8.
  For non-LM bifurcation lesion involving the MSA should be ≥6 mm2 in the main vessel; and the MSA in the ostial side branch should be ≥5 mm2 and ≥90% of distal reference lumen area; and symmetry index should be >0.8.
  Interventions: Procedure: Stenting
- Angiography-guided DK crush stenting (Active Comparator): In the Angiography-guided DK crush stenting group, stent diameter and length will be selected by visual estimation with a stent/artery ratio of 1.1:1.0. Post-dilation with a noncompliant balloon (balloon/stent diameter=1.0:1.0) inflated at >18 atm will be performed for all lesions. Angiographic success is defined as Thrombolysis In Myocardial Infarction (TIMI) grade 3, residual stenosis <20%, and the absence of ≥Type B dissection.
  Interventions: Procedure: Stenting

INTERVENTIONS:
Procedure: Stenting — DK crush technique with SYNERGY (Boston Scientific) drug-eluting stent implantation.

SUMMARY:
This study is designed to investigate whether IVUS-guided DK crush stenting technique compared to angiography-guided DK crush after the indexed procedure will lead to lower rates of the composite endpoint of target vessel failure (TVF) at 12 months. The individual components of TVF include cardiac death, target-vessel myocardial infarction (MI), or target vessel revascularization (TVR). Complex bifurcation lesions were defined according to DEFINITION study.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized-controlled, single blind, superiority trial that will include 35 international sites. The investigators aim to enroll 556 subjects with complex coronary bifurcation lesions in native coronary arterial segments.

All patients with complex coronary bifurcation lesions suitable for DES implantation will undergo 1:1 randomization either to IVUS-guided or angiography-guided DK crush stenting using a randomization schedule blocked by site.

All subjects will be screened according to the predefined inclusion and exclusion criteria per protocol and will further undergo angiography before DES implantation. Data and images will be collected during the index procedure, during re-intervention in the case of clinically driven TVF, and at the predefined 12-month clinical follow-up visit. All subjects will also undergo angiographic follow-up at 13 months.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures;
2. Men and women 18 years and older;
3. Established indication for PCI according to the guidelines of ACC/AHA;
4. Native coronary lesion suitable for drug-eluting stent placement;
5. True bifurcation lesions (Medina 0,1,1/1,1,1), lesions length≤ 68 mm
6. Reference vessel diameter in side branch > 2.5mm by visual estimation;
7. Complex bifurcation lesions based on the DEFINITION study.

Exclusion Criteria:

1. Pregnancy and breast feeding mother;
2. Co-morbidity with an estimated life expectancy of < 50 % at 12 months;
3. Scheduled surgery interrupting antiplatelet medications in the next 6 months;
4. Intolerable to DAPT;
5. Inability to follow the protocol and comply with follow-up requirements or any other reason that the investigator feels would place the patient at increased risk;
6. Unable to provide written informed consent, or fail to follow the protocol;
7. Previous enrolment in coronary intervention device investigation during the study period;
8. Lesion cannot be covered by 2 longest stents;
9. Restenotic bifurcation lesions；
10. Severe calcification requiring rotational atherectomy;
11. Acute myocardial infarction less than 24 hours;
12. Chronic total occlusion which is not recanalized;
13. Simple bifurcation lesions;
14. Renal failure requiring or during dialysis;
15. Hemoglobin <9g/L
16. Uncontrolled hypertension (systolic blood pressure≥180 mmHg or diastolic blood pressure≥110 mmHg)
17. Severe heart failure (LVEF<30%)
18. Combined pre- and post-capillary hypertension (mPAP≥25 mmHg, PCWP>15 mmHg, and PVR>3.0 WU)
19. Patients with hypertrophic obstructive cardiomyopathy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 556 (Actual)
Dates: Start 2018-12-26 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of target vessel failure | 12 months after DES implantation
  TVF defined as the composite of cardiac death, target vessel myocardial infarction (TVMI), and clinically driven TVR.

SECONDARY OUTCOMES:
Rate of stent thrombosis | 12 months after DES implantation
  The safety endpoint was stent thrombosis (ST), according to the definition by Academic Research Consortium.

CONTACTS AND LOCATIONS:
Overall Officials: Shao-Liang Chen, MD, PhD, Study Chair — Nanjing First Hospital, Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen SL, Sheiban I, Xu B, Jepson N, Paiboon C, Zhang JJ, Ye F, Sansoto T, Kwan TW, Lee M, Han YL, Lv SZ, Wen SY, Zhang Q, Wang HC, Jiang TM, Wang Y, Chen LL, Tian NL, Cao F, Qiu CG, Zhang YJ, Leon MB. Impact of the complexity of bifurcation lesions treated with drug-eluting stents: the DEFINITION study (Definitions and impact of complEx biFurcation lesIons on clinical outcomes after percutaNeous coronary IntervenTIOn using drug-eluting steNts). JACC Cardiovasc Interv. 2014 Nov;7(11):1266-76. doi: 10.1016/j.jcin.2014.04.026. Epub 2014 Oct 15. PMID 25326748
- [Derived] Ge Z, Kan J, Gao XF, Kong XQ, Zuo GF, Ye F, Tian NL, Lin S, Liu ZZ, Sun ZQ, He PC, Wei L, Yang W, He YQ, Xue YZ, Wang LM, Miao LF, Pu J, Sun YW, Nie SP, Tao JH, Wen SY, Yang Q, Su X, Yao QC, Huang YJ, Xia Y, Shen FR, Qiu CG, Mao YL, Liu Q, Hu XQ, Du ZM, Nie RQ, Han YL, Zhang JJ, Chen SL. Comparison of intravascular ultrasound-guided with angiography-guided double kissing crush stenting for patients with complex coronary bifurcation lesions: Rationale and design of a prospective, randomized, and multicenter DKCRUSH VIII trial. Am Heart J. 2021 Apr;234:101-110. doi: 10.1016/j.ahj.2021.01.011. Epub 2021 Jan 16. PMID 33465369